CLINICAL TRIAL: NCT06406426
Title: An Open and Exploratory Study of The Second-line Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma With Cadonilimab and Fruquintinib Combined With Paclitaxel-albumin
Brief Title: Study of The Second-line Treatment of Advanced Gastric / Gastroesophageal Junction Adenocarcinoma With Cadonilimab and Fruquintinib Combined With Paclitaxel-albumin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Director of Department of Medical Oncology, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFPG2024
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gastric / Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who have failed previous standard chemotherapy in the first line (Experimental)
  Interventions: Drug: Cadonilimab and Fruquintinib Combined With Paclitaxel-albumin
- Patients who had failed PD-1/L1 antibody combined chemotherapy in the first line (Experimental)
  Interventions: Drug: Cadonilimab and Fruquintinib Combined With Paclitaxel-albumin

INTERVENTIONS:
Drug: Cadonilimab and Fruquintinib Combined With Paclitaxel-albumin — Cadonilimab : 6mg/kg (≤375mg) d1,15 s.c. Q4W; Fruquintinib: 3mg p.o. Q.d d1-21,Q4W.; Paclitaxel-albumin: 100 mg/m2 d1,8,15 stop for one week, i.v. Q4W

SUMMARY:
This study is a prospective, open-label, two-arm exploratory Phase II clinical trial aimed at observing and evaluating the efficacy and safety of combined therapy with cadonilimab and fruquintinib in conjunction with paclitaxel-albumin as second-line treatment for advanced gastric/esophagogastric junction adenocarcinoma. Patients meeting the inclusion criteria were divided into two groups based on whether they had received PD-1/L1 antibody treatment in the first line: Group A (immunotherapy-naive group - patients who had previously failed standard chemotherapy in the first line) and Group B (immunotherapy rechallenge group - patients who had previously failed PD-1/L1 antibody combined chemotherapy in the first line). All patients received combined therapy with cadonilimab and fruquintinib in conjunction with paclitaxel-albumin until intolerable toxic reactions occurred, disease progression, withdrawal of informed consent by the subject, loss to follow-up, death, other conditions judged by the investigator to require termination of treatment, or termination of the study, whichever occurred first. The maximum duration of paclitaxel-albumin treatment was 6 cycles, and cadonilimab treatment did not exceed 1 year. Clinical tumor imaging evaluations were conducted every 8 weeks during treatment using RECIST v1.1 criteria, and safety assessments were performed using CTCAE 5.0, recording adverse events within 30 days from the first dose to the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent prior to enrollment. Age 18-80 years. Negative for HER2 Diagnosis confirmed by histological examination and/or cytological examination combined with imaging assessment of advanced metastatic gastric/gastroesophageal junction adenocarcinoma.

Failure of previous first-line therapy. Group A (immunotherapy naive ): patients who have failed prior chemotherapy with first-line standard therapy. Group B (immunotherapy rechallenge): patients who had previously failed PD-1/L1 antibody combined chemotherapy in the first line.

ECOG score: 0 to 1. At least one measurable lesion (≥10 mm long diameter on CT scan for non-lymph node lesions and ≥15 mm short diameter on CT scan for lymph node lesions according to iRECIST criteria).

Adequate organ function with. Routine blood: Absolute Neutrophil Count (ANC) 1.5 × 109/L, Platelets (Platelet, PLT) ≥ 100 × 109/L, Hemoglobin (HGB) ≥ 90 g/L.

Liver function: Total Bilirubin (TBIL) ≤ 1.5 × Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤3×ULN; serum albumin ≥30 g/L; after conventional hepatoprotective treatment meeting the above criteria, and can be stable for at least 1 week after evaluation by the investigator can be enrolled.

Renal function: Creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/mi (applying the standard Cockcroft-Gault formula).

Coagulation function: International Normalized Ratio (INR) ≤ 1.5 /PT ≤ 1.5 × ULN, aPTT ≤ 1.5 × ULN; if the subject is receiving anticoagulation therapy, as long as PT and INR are within the range drawn up by anticoagulant drugs.

A predicted survival of ≥ 3 months. Female patients must be non-pregnant and non-lactating and are required to use a medically approved form of contraception (e.g., IUD, pill or condom) during study treatment and for at least 120 days after study completion, and are not allowed to donate eggs to another person or freeze them for fertilization and propagation during this period.

Exclusion Criteria:

Symptomatic brain metastases. Known MSI-H/dMMR. A prior history of a primary tumor outside of the gastric/gastroesophageal junction in 3 years Active autoimmune disease or autoimmune disease with potential for recurrence such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, previous thyroid surgery cannot be included; subjects with vitiligo or complete remission of asthma in childhood and adult who do not require any intervention afterwards can be included; subjects with asthma requiring medical intervention with bronchodilators cannot be included.

Subjects with any severe and/or uncontrolled disease. including. Poorly controlled blood pressure (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); poorly controlled diabetes (fasting blood glucose [FBG] > 10 mmol/L) Having ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470ms) and ≥ grade 2 congestive heart failure (New York Heart Association [NYHA] classification) Active or uncontrolled severe infection (≥ CTCAE grade 2 infection) requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection Active hepatitis (transaminases do not meet the inclusion criteria, hepatitis B reference: HBV DNA ≥ 1000 IU/ml or ≥ 10^4 copies/ml; hepatitis C reference: HCV RNA ≥ 1000 IU/ml or ≥ 10^4 copies/ml; after nucleotide based antiviral therapy below the above criteria, can be enrolled); chronic hepatitis B virus carriers with HBV DNA < 10^4 IU/ml, who must receive concomitant antiviral therapy during the trial to be enrolled.

Those with renal failure requiring hemodialysis or peritoneal dialysis. Those with a history of immunodeficiency, including HIV-positive or suffering from other acquired or congenital immunodeficiency diseases, or a history of organ transplantation Active autoimmune disease requiring systemic therapy (e.g., use of disease-relieving drugs, corticosteroids, or immunosuppressive agents) within 2 years prior to the start of study treatment, except for replacement therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency); receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy. Doses >10 mg/day of prednisone or other equivalent hormone and within 2 weeks of the first dose and still continuing Those with a history of active tuberculosis Those who fail to control and still require repeated drainage of ascites, pericardial effusion, pleural effusion.

Research treatment related to. Patients who have undergone major organ transplantation Those who have undergone major surgical treatment, incisional biopsy or significant traumatic injury within 28 days prior to the start of study treatment; or have a long-standing untreated wound or fracture History of live attenuated vaccination within 14 days prior to the start of study treatment or planned live attenuated vaccination during the study History of severe hypersensitivity reactions following the use of monoclonal antibodies; known hypersensitivity to active ingredients or excipients such as envafolimab, lenvatinib, etc., of this study drug Those who are participating or have participated in other clinical studies within 4 weeks prior to the start of the study Those who have received taxanes, anti-angiogenic agents, and dual immunotherapy during first-line treatment.

Those with a history of severe allergy. Women who are pregnant or breastfeeding At risk for bleeding, or with coagulation disorders, or undergoing thrombolytic therapy Those with a history of psychotropic substance abuse and unable to abstain or with psychiatric disorders Subjects who, in the judgment of the investigator, have a concomitant disease that seriously jeopardizes the safety of the subject or interferes with the completion of the study, or subjects for whom other reasons are deemed to exist that make them unsuitable for enrollment In the judgment of the investigator, subjects who, in the judgment of the investigator, have a concomitant disease that seriously jeopardizes the safety of the subject or interferes with the completion of the study, or subjects for whom other reasons are deemed to exist that make them unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with measurable lesions achieving a Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) criteria.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 12 months
  Time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.
Disease Control Rate (DCR) | 12 months
  The proportion of participants who achieves a best overall response of CR, PR or stable disease(SD).
Duration of Response (DoR) | 12 months
  The time from the date that response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Overall Survival (OS) | 18months
  OS is defined as the time from enrollment to death from any cause.
Adverse Events (AEs) | [Time Frame: 12 months]
  Adverse Events (AEs) according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No